CLINICAL TRIAL: NCT03702153
Title: The Use of Synthetic Mesh in Contaminated and Infected Abdominal Wall Repairs: Challenging the Dogma of an Absolute Contra-indication. A Long-term Prospective Clinical Trial
Brief Title: The Use of Synthetic Mesh in Contaminated and Infected Abdominal Wall Repairs. A Long-term Prospective Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Claudio Birolini, MD, PhD, University of Sao Paulo General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PPM - Prospective
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Abdominal Wall Defect; Abdominal Wall Infection; Abdominal Wall Fistula; Infection
Keywords: ventral hernia; mesh infection; enteric fistula; polypropylene mesh; synthetic mesh; abdominal wall reconstruction; complex hernia
MeSH Terms: conditions — Infections; Hernia, Ventral | interventions — Abdominoplasty

STUDY DESIGN:
Intervention Model Description: A study group submitted to abdominal wall repair with synthetic mesh in the contaminated/infected setting compared to a control group submitted to abdominal wall repair with synthetic mesh in the clean setting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infected abdominal wall group (Experimental): A cohort of 40 patients carrying an active chronic mesh infection (mesh sinus, exposed mesh or mesh related enteric fistulas) resulting from a previous hernia repair, with or without an associated recurrent ventral hernia, and submitted to abdominal wall reconstruction with synthetic mesh.
  Interventions: Procedure: Abdominal wall reconstruction
- Clean control group (Active Comparator): A cohort of 40 patients with ventral hernias, and submitted to clean ventral hernia repair with synthetic mesh.
  Interventions: Procedure: Abdominal wall reconstruction

INTERVENTIONS:
Procedure: Abdominal wall reconstruction — The repair of abdominal wall defects with polypropylene mesh
  Other Names: Ventral hernia repair

SUMMARY:
Background: Abdominal wall reconstruction in patients presenting with enteric fistulas and mesh infection is challenging. There is a consensus that synthetic mesh must be avoided in infected operations. The alternatives to using synthetic mesh, such as component separation techniques and biologic mesh, present disappointing results with expressive wound infection and hernia recurrence rates.

Methods: A prospective clinical trial designed to evaluate the short and the long-term outcomes of patients submitted to elective abdominal wall repair with synthetic mesh in the dirty-infected setting, and compared to a cohort of patients submitted to clean ventral hernia repairs.

DETAILED DESCRIPTION:
We designed a prospective study, evaluating the short and the long-term outcomes of the surgical treatment of 40 consecutive patients presenting with an infected abdominal wall, compared to a cohort of 40 patients submitted to clean ventral hernia repairs. Patients were admitted between January 2012 and February 2015, and operated at the Hospital das Clinicas of the University of São Paulo School of Medicine, in Brazil. All patients included in the study group carried an active chronic mesh infection (mesh sinus, exposed mesh or mesh related enteric fistulas) resulting from a previous hernia repair, with or without an associated recurrent ventral hernia. All the operations required in this group were classified as Class IV (dirty-infected), accordingly to the CDC Wound Classifications, as adopted by the European registry for abdominal wall hernias. The only inclusion criterion was the presence of an active chronic mesh infection. The infected abdominal wall (IM) group and the outcomes of the treatment were compared to a clean-control (CC) group of patients who underwent clean abdominal wall reconstructions, originally belonging to a prospective study of the tensiometry of the abdominal wall, and operated during the same period and in the same conditions. The exclusion criteria were: giant ventral hernias with a volume ratio higher than 25%, patients on immunosuppressive therapy or using corticosteroids, patients with hepatic cirrhosis and portal hypertension, Chron´s disease, acute postoperative mesh infection, chronic mesh infections following inguinal hernia repair and emergency operations.The data assessed included gender, age, body mass index (BMI), American Society of Anesthesiologists (ASA) score, comorbidities, smoking status, cancer history, the number of previous abdominal operations, the number of prior hernia operations, the presence of a recurrent incisional hernia and/or enteric fistula and the presentation of the mesh infection. Perioperative data included operative time, anesthesia time, associated procedures, the defect characteristics and the extension of the pre-aponeurotic dissection. Further analysis in the infected mesh (IM) group included the type and position of the infected mesh, the causes for the mesh infection and the microbiology of mesh explants. Patients were followed and operated at the Abdominal Wall and Hernia Repair Unit of the General Surgery and Trauma Discipline, and five surgeons of the team conducted the operations in both groups. Informed consents were presented to the patients in the IM group upon admission. Patients in the CC group signed informed consents to participate the study, during their post-operative follow-up visits.

Surgical procedure The operations were performed through the previous surgical incision. Patients in the IM group had the infected mesh removed completely together with all the sutures, tacks or other foreign material. The surrounding fibrotic tissue and the existing sinus tracts were resected to perform a complete toilet of the abdominal wall. The abdominal cavity was entered in most of the patients, and associated or incidental procedures were made as required. After the removal of the infected mesh, or at the end of the abdominal cavity workup, all the surgical drapes, instruments and gloves were replaced. The size of the defect and the extension of the anterior abdominal wall dissection were estimated. The reconstruction of the midline was done as anatomically as possible, by repositioning of the muscles and primary closure of the aponeurosis. We did not use component separation techniques or transverse abdominal releases in any case. In some patients, a bilateral relaxing incision along the anterior rectus sheath was required to allow the re-approximation of the muscles in the midline. In all patients, a heavyweight macroporous (pore size > 75µm) monofilament polypropylene mesh (Intracorp®, Venkuri, www.venkuri.com.br) was used in the onlay position, to reinforce the repair. The mesh was fixed with multiple absorbable Vicryl® sutures, placed over the borders of the mesh, in the midline and along the relaxing incisions. The remaining dead space between the mesh and the underlying tissue was cleared entirely with interrupted sutures. The operative field was irrigated with 0,9% saline, and the subcutaneous was drained with suction drains. The scars and the exceeding skin flaps were resected. We did not use irrigation with antibiotics solution. The subcutaneous tissue and the skin were closed with interrupted sutures. Fluids and samples of the explanted mesh were sent to cultures and microbiological analysis. The same technique of repair was used in the CC group. The size of the defect was measured, and the extension of the anterior abdominal wall dissection was estimated. A bilateral relaxing incision along the anterior rectus sheath was used routinely in this group, to allow a tensionless closure of the midline.

Outcomes parameters The primary outcomes variables were the presence of any surgical site occurrences (SSO) or surgical site infection (SSI) during the first 30 days after the operation, and the development of hernia recurrence or the recurrence of mesh infection during a 36-month follow-up period. Suspected recurrences of a hernia or infection were determined by physical examination and CT scan imaging. Non-surgical complications, other operations, and deaths were registered during the follow-up period.

Statistical Analysis The chi-square test was conducted to verify the association between categorical variables in contingency tables and the Fisher exact test was adopted in 2x2 tables whenever at least one expected frequency was less than 5. The U-test was used for verifying the association between continuous data and group with two categories, and when normal distribution was observed the Student t-test was performed. The 5% level of significance was considered for all statistical tests. Statistical computer Stata software version 10.0 (StataCorp, College Station, TX) was used for conducting all statistical analysis.

ELIGIBILITY:
"Inclusion Criterion"

- the presence of an active chronic mesh infection

"Exclusion Criteria"

* giant ventral hernias with a volume ratio higher than 25% and loss of domicile
* patients on immunosuppressive therapy or using corticosteroids
* patients with hepatic cirrhosis and portal hypertension
* Chron´s disease
* acute postoperative mesh infection
* chronic mesh infections following inguinal hernia repair
* emergency operations.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2015-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Surgical site occurrence | 30 days
  any surgical infection, wound breakdown, soft tissue ischemia, seroma and hematoma formation

SECONDARY OUTCOMES:
Surgical Site infection | 30 days
  an infection occurring in the part of the body where the surgery took place and further defined as superficial, deep, and organ space
Surgical site occurrence requiring procedural intervention | 30 days
  any wound event requiring opening of the wound, wound debridement, suture excision, percutaneous drainage, hematoma evacuation, or mesh removal
Ventral hernia recurrence | 36 months
  a recurrence of ventral hernia
Mesh infection recurrence | 36 months
  a recurrence of mesh infection

OTHER OUTCOMES:
Microbiology of mesh infection | 30 days
  a study of the microorganisms causing chronic mesh infection

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Birolini, MD, Principal Investigator — Hospital das Clínicas da FMUSP
Locations (1):
- Hospital das Clinicas da FMUSP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Brief records and pictures, both of the operations and follow up data, are available.
Supporting Information: CSR
Time Frame: From march 2018, available for 1 year
Access Criteria: Available data to be shared with researchers interested in abdominal wall reconstruction
URL: https://vimeo.com/90585364

REFERENCES:
- [Background] Choi JJ, Palaniappa NC, Dallas KB, Rudich TB, Colon MJ, Divino CM. Use of mesh during ventral hernia repair in clean-contaminated and contaminated cases: outcomes of 33,832 cases. Ann Surg. 2012 Jan;255(1):176-80. doi: 10.1097/SLA.0b013e31822518e6. PMID 21677561
- [Background] Szczerba SR, Dumanian GA. Definitive surgical treatment of infected or exposed ventral hernia mesh. Ann Surg. 2003 Mar;237(3):437-41. doi: 10.1097/01.SLA.0000055278.80458.D0. PMID 12616130
- [Background] Johnson EK, Tushoski PL. Abdominal wall reconstruction in patients with digestive tract fistulas. Clin Colon Rectal Surg. 2010 Sep;23(3):195-208. doi: 10.1055/s-0030-1262988. PMID 21886470
- [Background] Franklin ME Jr, Trevino JM, Portillo G, Vela I, Glass JL, Gonzalez JJ. The use of porcine small intestinal submucosa as a prosthetic material for laparoscopic hernia repair in infected and potentially contaminated fields: long-term follow-up. Surg Endosc. 2008 Sep;22(9):1941-6. doi: 10.1007/s00464-008-0005-y. Epub 2008 Jul 2. PMID 18594919
- [Background] Miserez M, Fitzgibbons RJ Jr, Schumpelick V. Hernia surgery and contamination: biological mesh and nothing else? Hernia. 2013 Feb;17(1):1. doi: 10.1007/s10029-013-1044-4. Epub 2013 Jan 17. No abstract available. PMID 23324870
- [Background] Itani KM, Rosen M, Vargo D, Awad SS, Denoto G 3rd, Butler CE; RICH Study Group. Prospective study of single-stage repair of contaminated hernias using a biologic porcine tissue matrix: the RICH Study. Surgery. 2012 Sep;152(3):498-505. doi: 10.1016/j.surg.2012.04.008. Epub 2012 Jul 3. PMID 22763262
- [Background] Rosen MJ, Denoto G, Itani KM, Butler C, Vargo D, Smiell J, Rutan R. Evaluation of surgical outcomes of retro-rectus versus intraperitoneal reinforcement with bio-prosthetic mesh in the repair of contaminated ventral hernias. Hernia. 2013 Feb;17(1):31-5. doi: 10.1007/s10029-012-0909-2. Epub 2012 Mar 14. PMID 22415440
- [Background] Rosen MJ, Krpata DM, Ermlich B, Blatnik JA. A 5-year clinical experience with single-staged repairs of infected and contaminated abdominal wall defects utilizing biologic mesh. Ann Surg. 2013 Jun;257(6):991-6. doi: 10.1097/SLA.0b013e3182849871. PMID 23426340
- [Background] Birolini C, Utiyama EM, Rodrigues AJ Jr, Birolini D. Elective colonic operation and prosthetic repair of incisional hernia: does contamination contraindicate abdominal wall prosthesis use? J Am Coll Surg. 2000 Oct;191(4):366-72. doi: 10.1016/s1072-7515(00)00703-1. PMID 11030241
- [Background] Antonopoulos IM, Nahas WC, Mazzucchi E, Piovesan AC, Birolini C, Lucon AM. Is polypropylene mesh safe and effective for repairing infected incisional hernia in renal transplant recipients? Urology. 2005 Oct;66(4):874-7. doi: 10.1016/j.urology.2005.04.072. PMID 16230159
- [Background] Birolini C, de Miranda JS, Utiyama EM, Rasslan S. A retrospective review and observations over a 16-year clinical experience on the surgical treatment of chronic mesh infection. What about replacing a synthetic mesh on the infected surgical field? Hernia. 2015 Apr;19(2):239-46. doi: 10.1007/s10029-014-1225-9. Epub 2014 Feb 9. PMID 24509890
- [Derived] Birolini C, Faro Junior MP, Terhoch CB, de Miranda JS, Tanaka EY, Utiyama EM. Microbiology of chronic mesh infection. Hernia. 2023 Aug;27(4):1017-1023. doi: 10.1007/s10029-023-02747-6. Epub 2023 Feb 9. PMID 36757611
- [Derived] Birolini C, de Miranda JS, Tanaka EY, Utiyama EM, Rasslan S, Birolini D. The use of synthetic mesh in contaminated and infected abdominal wall repairs: challenging the dogma-A long-term prospective clinical trial. Hernia. 2020 Apr;24(2):307-323. doi: 10.1007/s10029-019-02035-2. Epub 2019 Sep 6. PMID 31493051